CLINICAL TRIAL: NCT06023095
Title: A Multiple Dose Titration Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3502970 in Chinese Participants Who Have Obesity or Are Overweight With Weight-related Comorbidities
Brief Title: A Study of LY3502970 in Chinese Participants With Obesity or Are Overweight With Weight-related Comorbidities
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18610; J2A-GH-GZGX (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Overweight; Obesity
Keywords: Safety and Tolerability; Chinese; LY3502970
MeSH Terms: conditions — Overweight; Obesity | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY3502970 (Experimental): LY3502970 administered orally
  Interventions: Drug: LY3502970
- Placebo (Placebo Comparator): Placebo administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3502970 — Administered orally.
  Arms: LY3502970
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn about the safety and tolerability of LY3502970 when given to Chinese participants with obesity or overweight with weight-related comorbidities. Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body. Each enrolled participant will receive LY3502970, or placebo given orally. For each participant, the study will last about approximately 22- and 30-weeks for both cohort 1 and 2, respectively including screening period.

ELIGIBILITY:
Inclusion Criteria:

* Are native Chinese males or females
* Have had a stable body weight for the 3 months prior to randomization (less than 5% body weight change) and body mass index of ≥ 30.0 kilograms per square meter (kg/m²) or between 27.0 up to 30.0 kg/m² with at least 1 of the following weight-related comorbidities including Hypertension, Dyslipidemia, Cardiovascular disease, Obstructive sleep apnea

Exclusion Criteria:

* Have any prior diagnosis of type 1 diabetes mellitus (T1DM) or type 2 diabetes mellitus (T2DM), or rare forms of diabetes mellitus
* Have used or intend to use any prescription or over-the-counter medications or traditional Chinese treatments within 3 months prior to screening, exception of medications for the treatment of concurrent medical conditions with a stable dose
* Have known allergies to GLP-1RAs, LY3502970, related compounds, any components of the formulation, or have a history of significant atopy
* Are overweight or have obesity induced by other endocrinological disorders, diagnosed monogenetic, or syndromic forms of obesity
* Have or plan to have a surgical, endoscopic or device-based treatment for obesity
* Have a history or presence of psychiatric disorder, a moderately severe or severe depression status, or a significantly risk for suicide
* Have a history of acute or chronic pancreatitis
* Have a known self or family history of multiple endocrine neoplasia type 2A or type 2B, thyroid C-cell hyperplasia, or medullary thyroid carcinoma
* Have other acute, chronic, or uncontrolled medical conditions, vital organ failure or abnormal laboratory value in the judgment of the investigator would make the participant inappropriate for entry into this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Week 18 (Cohort 1) & Week 26 (Cohort 2)
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3502970 | Predose on Day 1 up to 116 (Cohort 1) & 172 (Cohort 2) Days postdose
  PK: Cmax of LY3502970
PK: Area Under the Concentration Versus Time Curve From Time 0 to 24 hour Time Point (AUC0-24) of LY3502970 | Predose on Day 1 up to 116 (Cohort 1) & 172 (Cohort 2) Days postdose
  PK: AUC0-24 of LY3502970
Pharmacodynamics (PD): Change From Baseline in Body Weight | Baseline through 113 Days (Cohort 1) and 169 Days (Cohort 2)
  PD: Change From Baseline in Body Weight
PD: Change From Baseline in Body Mass Index | Baseline through 113 Days (Cohort 1) and 169 Days (Cohort 2)
  PD: Change From Baseline in Body Mass Index
PD: Change From Baseline in Waist Circumference | Baseline through 113 Days (Cohort 1) and 169 Days (Cohort 2)
  PD: Change From Baseline in Waist Circumference
PD: Change From Baseline in Fasting Plasma Glucose | Baseline through 113 Days (Cohort 1) and 169 Days (Cohort 2)
  PD: Change From Baseline in Fasting Plasma Glucose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- China (3):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Shanghai General Hospital, Shanghai, Songjiang

IPD SHARING:
Plan to Share IPD: No